CLINICAL TRIAL: NCT02436122
Title: Prospective Cohort Study for the Impact of Preoperative Glycemic Control Status Measured by HbA1c Levels on Pathologic Features and Oncological Outcomes in the Patients With Prostate Cancer
Brief Title: Impact of Preoperative HbA1c Levels on Pathologic Features and Oncological Outcomes in the Patients With Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Kyu Hong, Associate professor, Seoul National University Hospital
Other Study IDs: B-1504-293
Record Dates: First submitted 2015-05-03; First posted 2015-05-06 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Neoplasm; Pathology
Keywords: Prostate cancer; Preoperative; Glycemic control; Hemoglobin A1c; Pathologic outcomes; Oncological outcomes; Treatment Outcome; Hemoglobin A1c Protein, Human
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The effect of preoperative glycemic control measured by HbA1c on prostate cancer (PCa) outcome remains controversial. Thus, the investigators aim to examine the association of preoperative glycemic control with oncologic outcomes after radical prostatectomy (RP).

The investigators will prospectively collect the relevant data including preoperative HbA1c in 264 patients of PCa patients undergoing RP. The associations between clinical variables and risk of adverse pathological features and disease recurrence will be tested using a multivariate logistic regression and multiple Cox-proportional hazards model, respectively.

DETAILED DESCRIPTION:
* This is the observational study as the single institutional, prospective cohort study. The investigators prospectively collect the clinicopathological information of the patients with prostate cancer (PCa) undergoing radical prostatectomy (RP).
* Particularly, the investigators check the variables, including age at surgery, body mass index, comorbidities, preoperative PSA levels, prostate volume measured by TRUS, preoperative HbA1c levels, biopsy Gleason score, positive biopsy cores, percent positive cores, clinical TMN staging, final pathological results (TMN stage, Gleason score, extraprostatic extension, seminal vesicle invasion, surgical margin positivity, postoperative biochemical recurrence (BCR), local recurrence, and distant metastasis during follow-up periods.
* The study protocol is same with routine follow-up schedule of the patients with PCa treated with RP. Typically, the investigators check the patients at 1, 3, 6, 9, 12, 18, 24, 30 and 36 months. However, according to the patients status and preference, follow-up schedule can be changed within 3 months at specific time points. Because the present study is the observational cohort study, not intervention study, subtle changes of follow-up schedule would not affect on the primary outcomes.
* Importantly, preoperative HbA1c should be checked within 1 month before operation, same as the routine preoperative laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer diagnosed with prostate biopsy
* Clinically localized PCa confirmed by prostate MRI and Bone scan
* Patients undergoing RP

Exclusion Criteria:

* Distant metastasis, preoperatively
* Preoperative hormone therapy
* Preoperative chemotherapy
* Radiation therapy
* Medications affecting glucose status other than diabetes mellitus

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled patients should be diagnosed with prostate cancer by TRUS-guided 12 cores biopsy. In addition, the participants should be treated with radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence (BCR) | postoperative up to 3 years
  BCR was defined as either two consecutive increases in serum PSA (>0.2 ng/mL) or the administration of adjuvant therapy during the postoperative follow-up period
Pathological Gleason score | within 2 weeks after surgery
  Gleason scores of prostate cancer specimen described in final pathological report

SECONDARY OUTCOMES:
Pathological TMN stage | within 2 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea